CLINICAL TRIAL: NCT02057991
Title: A Mindfulness-Based Educational Intervention For Colorectal Cancer Patients And Caregivers
Brief Title: Mindfulness-Based Exercise Video in Educating Hispanic/Latino Patients With Colorectal Cancer and Their Caregivers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient Accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3C-13-6; NCI-2014-00164 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 3C-13-6 (Other: USC Norris Comprehensive Cancer Center); R01CA155101 (NIH); P30CA014089 (NIH)
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Anxiety Disorder; Colon Cancer; Depression; Fatigue; Rectal Cancer
MeSH Terms: conditions — Anxiety Disorders; Colonic Neoplasms; Depression; Fatigue; Rectal Neoplasms | interventions — Early Intervention, Educational; Methods; Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group I (standard of care) (No Intervention): Patients and caregivers receive standard of care.
- Group II (educational video) (Experimental): Patients and caregivers receive a 20-minute self-playing interactive educational video brochure.
  Interventions: Other: educational intervention; Other: caregiver-related intervention or procedure; Other: questionnaire administration; Other: laboratory biomarker analysis
- Group III (educational video, mindfulness exercise video) (Experimental): Patients and caregivers receive a 20-minute self-playing interactive educational video brochure and watch a 20-minute interactive mindfulness exercise video.
  Interventions: Other: educational intervention; Procedure: CAM exercise therapy; Other: caregiver-related intervention or procedure; Other: questionnaire administration; Other: laboratory biomarker analysis

INTERVENTIONS:
Other: educational intervention — Watch an educational video
  Other Names: intervention, educational
  Arms: Group II (educational video); Group III (educational video, mindfulness exercise video)
Procedure: CAM exercise therapy — Watch a mindfulness exercise video
  Other Names: Exercise Therapy
  Arms: Group III (educational video, mindfulness exercise video)
Other: caregiver-related intervention or procedure — Watch mindfulness exercise video and/or educational video
  Arms: Group II (educational video); Group III (educational video, mindfulness exercise video)
Other: questionnaire administration — Ancillary studies
  Arms: Group II (educational video); Group III (educational video, mindfulness exercise video)
Other: laboratory biomarker analysis — Correlative studies
  Arms: Group II (educational video); Group III (educational video, mindfulness exercise video)

SUMMARY:
This randomized pilot trial studies mindfulness-based program in educating patients with colorectal cancer and their caregivers. A mindfulness-based exercise video may help reduce stress and fatigue in patients with colorectal cancer and their caregivers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effect of a brief educational program on colorectal cancer knowledge acquisition in a 3-arm randomized clinical trial (Control Group: standard of care; Treatment Group 1: cancer education; Treatment Group 2: mindfulness + cancer education) comparing visual/written educational material with and without mindfulness training to the standard of care.

II. To determine the priming effect of a brief mindfulness training on retaining knowledge of colorectal cancer education.

III. To determine the joint effect of colorectal cancer education delivered to both the patient and a caregiver on the overall colorectal cancer knowledge.

SECONDARY OBJECTIVES:

I. To examine the relative changes in psychobiological variables (stress, anxiety, depression, mindfulness, fatigue, life benefit) from pre (T0) to post (T1) intervention in the 3 arms of the clinical trials.

II. To measure changes in salivary cortisol levels as an indicator of acute stress reactivity across 4 time points across a one-hour period (i.e., 0 min, 20 min, 40 min, 60 min) during active chemotherapy (T1).

III. To determine the moderating effect of baseline peripheral levels of inflammation (interleukin-1 [IL-1], IL-6, c-reactive protein [CRP] and tumor necrosis factor alpha [TNFa]) on the trajectory of salivary cortisol reactivity.

OUTLINE: Patients and caregivers are randomized to 1 of 3 groups.

GROUP I: Patients and caregivers receive standard of care.

GROUP II: Patients and caregivers receive a 20-minute self-playing interactive educational video brochure.

GROUP III: Patients and caregivers receive a 20-minute self-playing interactive educational video brochure and watch a 20-minute interactive mindfulness exercise video.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with colorectal cancer
* Patients with at least one more chemotherapy appointment at the time of enrollment
* if patients have a caregiver, patients should agree to bring a caregiver to one of their hospital visits or have the caregiver schedule a separate study visit
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Illiterate participants
* Deaf participants
* Participants that do not read speak or understand either Spanish or English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2014-01-07 (Actual); Primary Completion 2016-11-09 (Actual); Study Completion 2017-11-09 (Actual)

PRIMARY OUTCOMES:
Change in self-reported stress levels assessed using pre- and post-test assessments | Baseline to up to 60 minutes
  The intervention effects will be examined using multi-level modeling (MLM). These analyses will include chi-square, t-tests, and one way analyses of variance (ANOVAs).
Change in colorectal cancer knowledge assessed using pre- and post-test assessments | Baseline to up to 60 minutes
  The intervention effects will be examined using multi-level modeling (MLM). These analyses will include chi-square, t-tests, and one way ANOVAs.

SECONDARY OUTCOMES:
Changes in salivary cortisol levels using chemiluminescence immunoassay | Baseline to up 60 minutes
  Cortisol slopes will be calculated with two distinct areas under the curve analyses using the trapezoid formula as outlined by Pruessner 2003. Data values will be entered into a two factor (group by time) multilevel MIXED linear regression model to calculate differences between the three groups. A Scheffe post hoc test will be employed to determine the direction of the differences between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Figueiredo, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States